CLINICAL TRIAL: NCT06525142
Title: The Effectiveness of Audiovisual Intervention on the Parent-Child Bonding, Parental Role Perception, and Well-Being in Fathers of Premature Infants
Brief Title: The Effectiveness of Audiovisual Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Li Yi-Chun, Neonatal intensive care nurse, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Li Yi-Chun
Record Dates: First submitted 2024-07-07; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Parent-Child Relations; Premature; Infant, Light-for-dates; Premature Infant Disease
Keywords: Parent-Child Bonding,Parental Role Perception,Well-Being
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: The investigators will compare the pre- and post-test methods bwtween the experimental groups and the control group. The fathers of enrolled preterm infants will fill in the structured questionnaires at the time before the intervention (Baseline data) and one month later after the intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Effectiveness of Audiovisual Intervention (Experimental): The study is to understand the current status of parent-child bond, parenting role perception and well-being of fathers of preterm infants, and to explore the effect of audio-visual interventions on parent-child bonding, parenting role perception and well-being of fathers of preterm infants
  Interventions: Behavioral: Audiovisual Intervention
- control (Placebo Comparator): The study is to understand the current status of parent-child bond, parenting role perception and well-being of fathers of preterm infants, and to explore the effect of audio-visual interventions on parent-child bonding, parenting role perception and well-being of fathers of preterm infants
  Interventions: Behavioral: Audiovisual Intervention

INTERVENTIONS:
Behavioral: Audiovisual Intervention — 【Group 1】During the first three days, the researchers will provide a storybook to the father of the premature infant, and the researchers assist in recording the father's voice of the storybook in the form of MP4 recording. At the fourth day, one hour after the baby feeding, the father's voice will be played by the player to the baby, for 2 consecutive days, 2 times/day, 10 minutes/time. The baby's heartbeat, breathing and blood oxygen changes will be recorded and monitored with a physiological monitor. The recording files will be kept by the researcher.
  【Group 2】 The intervention will be the same with Group 1 except the following intervention: on the 4th-6th day of the baby's birth, sleeping in the incubator, the baby's reaction behavior will be taken with a mobile phone, 1 time/day, 5 minutes/time, for 3 consecutive days, the image feedback is delivered to the father in person.

SUMMARY:
The objective of this clinical study is to understand the current status of parent-child bond, parenting role perception and well-being of fathers of preterm infants, and to explore the effect of audio-visual interventions on parent-child bonding, parenting role perception and well-being of fathers of preterm infants. The main questions it aims to answer are:

* After intervention, whether the parent-child connection between fathers and preterm infants in the audio-visual group is higher than that in the audio-visual group and the control group
* After the intervention, whether the father's perception of parenting role in the audio-visual group is higher than that of the vocal group and the control group
* After intervention, whether the father's happiness in the audio-visual group is higher than that in the audio-visual group and the control group The investigators will compare the pre- and post-test methods bwtween the experimental groups and the control group. The fathers of enrolled preterm infants will fill in the structured questionnaires at the time before the intervention (Baseline data) and one month later after the intervention.

DETAILED DESCRIPTION:
This study is a randomized controlled trial, which will compare the pre- and post-test methods between the experimental groups (2 groups) and the control group in an attempt to explore the effect of audio-visual intervention on the parent-child bond, parent-role perception and well-being of fathers of preterm infants.

The total number of participants is estimated as 99. All fathers of preterm infants will complete three questionnaires at the time of 1-3 days , one week, and one month of age of their preterm babies). It will take about 10-20 minutes for questionnaire survey each time. Study participants were randomly assigned to the following three groups (33 in each group):

【Group 1】During the first three days, the researchers will provide a storybook to the father of the premature infant, and the researchers assist in recording the father's voice of the storybook in the form of MP4 recording. At the fourth day, one hour after the baby feeding, the father's voice will be played by the player to the baby, for 2 consecutive days, 2 times/day, 10 minutes/time. The baby's heartbeat, breathing and blood oxygen changes will be recorded and monitored with a physiological monitor. The recording files will be kept by the researcher.

【Group 2】 The intervention will be the same with Group 1 except the following intervention: on the 4th-6th day of the baby's birth, sleeping in the incubator, the baby's reaction behavior will be taken with a mobile phone, 1 time/day, 5 minutes/time, for 3 consecutive days, the image feedback is delivered to the father in person.

【Group 3】This group is a control group. The fathers and preterm infants will not receive interventions conducted in group 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* father age > 20
* premature infant born at 29-36 weeks

Exclusion Criteria:

* infant failing the hearing examination
* father and mother are not married

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-06-04 (Estimated); Study Completion 2026-06-05 (Estimated)

PRIMARY OUTCOMES:
Postpartum Bonding Questionnaire | one month
  This questionnaire was designed by Brockington et al and published in 2001. The scale is a 5-point Likert's score. The higher score means a better parent-child bounding.
Paternal Role Significance Questionnaire | one month
  This questionnaire was designed by Bruce et al and published in 1999. The scale is a 4-point Likert's score. The higher score means a better significance of paternal role.
Satisfaction With Life Scale | one month
  This questionnaire was designed by Diener et al and published in 1985. The scale is a 7-point Likert's score. The higher score means a better satisfaction with life.
Positive and Negative Affect Schedule (PANAS) | one month
  This questionnaire was designed by Diener et al and published in 1995. The scale is a 7-point Likert's score. The higher score means more perceived happiness in life.

CONTACTS AND LOCATIONS:
Overall Officials: Hsing-Yi Yu,, Principal Investigator — Chang Gung University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Provenzi L, Broso S, Montirosso R. Do mothers sound good? A systematic review of the effects of maternal voice exposure on preterm infants' development. Neurosci Biobehav Rev. 2018 May;88:42-50. doi: 10.1016/j.neubiorev.2018.03.009. Epub 2018 Mar 10. PMID 29535067
- [Result] Rossen L, Hutchinson D, Wilson J, Burns L, A Olsson C, Allsop S, J Elliott E, Jacobs S, Macdonald JA, Mattick RP. Predictors of postnatal mother-infant bonding: the role of antenatal bonding, maternal substance use and mental health. Arch Womens Ment Health. 2016 Aug;19(4):609-22. doi: 10.1007/s00737-016-0602-z. Epub 2016 Feb 11. PMID 26867547
- [Result] Rowe HJ, Wynter KH, Steele A, Fisher JR, Quinlivan JA. The growth of maternal-fetal emotional attachment in pregnant adolescents: a prospective cohort study. J Pediatr Adolesc Gynecol. 2013 Dec;26(6):327-33. doi: 10.1016/j.jpag.2013.06.009. Epub 2013 Sep 26. PMID 24075091
- [Result] Sajjadian N, Mohammadzadeh M, Alizadeh Taheri P, Shariat M. Positive effects of low intensity recorded maternal voice on physiologic reactions in premature infants. Infant Behav Dev. 2017 Feb;46:59-66. doi: 10.1016/j.infbeh.2016.11.009. Epub 2016 Nov 30. PMID 27914263
- [Result] Makela H, Axelin A, Feeley N, Niela-Vilen H. Clinging to closeness: The parental view on developing a close bond with their infants in a NICU. Midwifery. 2018 Jul;62:183-188. doi: 10.1016/j.midw.2018.04.003. Epub 2018 Apr 11. PMID 29684798